CLINICAL TRIAL: NCT05533112
Title: Binaural Beat Stimulation as a Cost-effective Tool to Reduce Preoperative Anxiety and Improve Postoperative Outcome After General Anesthesia
Brief Title: Binaural Beat Stimulation to Improve Patient Outcome After Surgery and Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-332-S-NP
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Preoperative Anxiety; Perioperative Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Control Group, no Intervention received
- Preop Stimulation (Experimental): Binaural Beat Stimulation preoperatively
  Interventions: Other: Binaural Beat Stimulation
- Postop Stimulation (Experimental): Binaural Beat Stimulation postoperatively
  Interventions: Other: Binaural Beat Stimulation
- Pre- & Postop Stimulation (Experimental): Binaural Beat Stimulation pre- and postoperatively
  Interventions: Other: Binaural Beat Stimulation

INTERVENTIONS:
Other: Binaural Beat Stimulation — During binaural beats stimulation both ears receive a tone which varies slightly in its frequency. If the left ear is stimulated with a sinusoidal wave of 98 Hz and the right ear with a sinusoidal wave of 108 Hz, the brain will perceive this stimulation as a single tone at the mean frequency of 103 Hz. The amplitude of the perceived tone will fluctuate with a frequency that is equal to the difference of the two initial tones, i.e., 10 Hz
  Arms: Postop Stimulation; Pre- & Postop Stimulation; Preop Stimulation

SUMMARY:
We plan to evaluate the potential of binaural beat stimulation as a cost-effective tool to improve perioperative patient outcome. Preoperative anxiety and postoperative neurocognitive disorders are two major issues patients have to deal with in the perioperative period. In this context, preoperative stress and anxiety are independent risk factors for postoperative neurocognitive disorders. The primary goal of our proposed study therefore is to reduce preoperative anxiety by stimulating patients with binaural beats. As binaural beats might also entrain brainwaves, the secondary goal of the study is to investigate whether binaural beats can induce alpha oscillatory activity during emergence from anesthesia. This type of oscillation has been demonstrated to be protective for postoperative neurocognitive disorders and might therefore complement the effects of preoperative anxiety reduction.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in German (Munich) or Portuguese (Porto)
* Scheduled for elective minor or intermediate risk procedure

Exclusion Criteria:

* ASA status 4
* History of drug abuse
* Pre-existing neurocognitive or psychiatric disorders
* Auditory Impairments, vision diseases or other diagnosed cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of preoperative anxiety | Assessments will take place one day before surgery as well as before administration of the intervention
  Binaural beat stimulation before surgery can reduce preoperative anxiety

SECONDARY OUTCOMES:
Increase of EEG alpha-band power during anesthesia emergence | Analysis will include the last 20 minutes of surgical procedure until patients are responsive again
  Binaural beat stimulation during anesthesia emergence can increase or stabilize EEG alpha-band power.
Lower incidence of perioperative neurocognitive disorders | Incidence of perioperative neurocognitive disorders will be assessed during the patients stay in the PACU as well as one day post surgery
  2. Reduced preoperative anxiety and/or increased or stabilized alpha oscillations during anesthesia emergence are correlated with a lower incidence of perioperative neurocognitive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Kratzer, Dr., Principal Investigator — Klinik für Anästhesiologie und Intensivmedizin; Gerhard Schneider, Prof., Study Chair — Klinik für Anästhesiologie und Intensivmedizin; Matthias Kreuzer, Dr., Principal Investigator — Klinik für Anästhesiologie und Intensivmedizin
Locations (1):
- Technische Universität München, München, München (Stadt), Germany

IPD SHARING:
Plan to Share IPD: Yes
All recorded data may be shared with collaborating researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting March 2023.
Access Criteria: Researchers who agree to collaborate on the project will have access to our protected server and can access all recorded data.